CLINICAL TRIAL: NCT00974259
Title: Phase 2, Randomized Clinical Trial of the Safety and Efficacy of Brain Tissue Oxygen Monitoring in the Management of Severe Traumatic Brain Injury.
Brief Title: Brain Tissue Oxygen Monitoring in Traumatic Brain Injury (TBI)
Acronym: BOOST 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Washington (Other); University of Miami (Other); University of Pittsburgh (Other); Duke University (Other); Ohio State University (Other); Temple University (Other); Thomas Jefferson University (Other); University of Cincinnati (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Ramon Diaz-Arrastia, Professor of Neurology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01NS061860 (NIH); R01NS061860 (NIH); R01NS061860-01A2 (NIH)
Record Dates: First submitted 2009-09-04; First posted 2009-09-10 (Estimated); Results first posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Severe Traumatic Brain Injury
Keywords: Hypoxia; Ischemia; Intracranial hypertension; Neurocritical care
MeSH Terms: conditions — Brain Injuries, Traumatic; Hypoxia; Ischemia; Intracranial Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- pBrO2 and ICP management (Experimental): Treatment protocol based on pBrO2 and ICP values.
  Interventions: Device: Management protocol based on pBrO2 and ICP values.
- ICP management (Active Comparator): Treatment protocol based on ICP values only.
  Interventions: Device: Management protocol based on ICP values only.

INTERVENTIONS:
Device: Management protocol based on pBrO2 and ICP values. — For patients who experience falls in pBrO2 below 20 mm Hg, a hierarchical treatment algorithm will be instituted, adapted from published recommendations49. In principle, episodes requiring therapy will fall into one of 4 scenarios (scenario A, B, C, and D, defined in figure 7), which will require different management strategies. The treatment protocol depends on which type of episode is being treated. Treatment is triggered by abnormalities in either ICP (> 20 mm Hg) or pBrO2 (< 20 mm Hg) are noted. Elevations in ICP above 20 mm Hg or decline in pBrO2 below 20 mm Hg for more than 5 minutes will trigger a treatment intervention. Treatment is directed to an episode. Patients may start in one type of episode and move to another. Therapy will depend on which type of episode they are in at any given time.
  Other Names: Licox; Camino
  Arms: pBrO2 and ICP management
Device: Management protocol based on ICP values only. — For the patients randomized to ICP treatment alone, only Scenario A and Scenario B episodes are relevant.
  Other Names: Camino
  Arms: ICP management

SUMMARY:
Traumatic brain injury (TBI) is a major cause of death and disability, with an estimated cost of 45 billion dollars a year in the United States alone. Every year, approximately 1.4 million sustain a TBI, of which 50,000 people die, and another 235,000 are hospitalized and survive the injury. As a result, 80,000-90,000 people experience permanent disability associated with TBI. This project is designed to determine whether a device designed to measure brain tissue oxygenation and thus detect brain ischemia while it is still potentially treatable shows promise in reducing the duration of brain ischemia, and to obtain information required to conduct a definitive clinical trial of efficacy.

A recently approved device makes it feasible to directly and continuously monitor the partial pressure of oxygen in brain tissue (pBrO2). Several observational studies indicate that episodes of low pBrO2 are common and are associated with a poor outcome, and that medical interventions are effective in improving pBrO2 in clinical practice. However, as there have been no randomized controlled trials carried out to determine whether pBrO2 monitoring results in improved outcome after severe TBI, use of this technology has not so far been widely adopted in neurosurgical intensive care units (ICUs). This study is the first randomized, controlled clinical trial of pBrO2 monitoring, and is designed to obtain data required for a definitive phase III study, such as efficacy of physiologic maneuvers aimed at treating pBrO2, and feasibility of standardizing a complex intensive care unit management protocol across multiple clinical sites.

Patients with severe TBI will be monitored with Intracranial pressure monitoring (ICP) and pBrO2 monitoring, and will be randomized to therapy based on ICP along (control group) or therapy based on ICP in addition to pBrO2 values (treatment group). 182 participants will be enrolled at four clinical sites, the University of Texas Southwestern Medical Center/Parkland Memorial Hospital, the University of Washington/Harborview Medical Center, the University of Miami/Jackson Memorial Hospital, and the University of Pennsylvania/Hospital of the University of Pennsylvania. Functional outcome will be assessed at 6-months after injury.

DETAILED DESCRIPTION:
Design and Outcomes

This study is a two-arm, single-blind, randomized, controlled, phase II, multi-center pilot trial of the efficacy of pBrO2 monitoring, and is designed to obtain data required for a definitive phase III study, such as efficacy of physiologic maneuvers aimed at normalizing pBrO2. 182 patients with severe TBI who require ICP monitoring will be recruited into this study at 4 clinical sites in the US (Univ. of Texas Southwestern/Parkland Memorial Hospital, Univ. of Washington/Harborview Medical Center, Univ. of Miami/Jackson Memorial Hospital, and Univ. of Pennsylvania/Hospital of the Univ. of Pennsylvania). All patients will have both ICP monitors and pBrO2 monitors inserted through the same burr hole. Half of the patients will be randomized to a treatment protocol based on both ICP and pBrO2 readings, while the control group will be randomized to a treatment protocol based only on ICP readings. The pBrO2monitors of the control arm will be masked, so that the treating physicians will be unaware of the pBrO2 information. Patients will have telephone follow-up interview to assess their level of recovery 6 months post injury, using the Glasgow Outcome Scale-Extended.

Interventions and Duration

Patients randomized to the control group will have pBrO2 implanted in a similar fashion as patients in the treatment group, but after calibration of the device, the display will be covered with opaque tape. Patients in the control will be treated with a protocol based on ICP measures only. Patients in the treatment group (both ICP and pBrO2 measures are visible) will be treated according to a protocol that incorporates both ICP and pBrO2 measures. The treatment protocols are based on current standards of care, but are described in detail to insure uniformity in treatments across the 4 study sites.

The probe will remain in place for a maximum or 5 days, until all values are normal for 48 hours, or sooner if a complication arises. If the patient has normal values, monitors will be removed after 48 hours.

Objectives

Primary Objective: The prescribed treatment protocol, based on pBrO2 monitoring, results in reduction of the fraction of time that brain oxygen levels are below the critical threshold of 20 mm Hg in patients with severe traumatic brain injury.

Secondary Objectives:

* Safety hypotheses: Adverse events associated with pBrO2 monitoring are rare.
* Feasibility hypotheses: Episodes of decreased pBrO2 can be identified and treatment protocol instituted comparably across 4 clinical sites, and protocol violations will be low (<10%) and uniform across different clinical sites.
* Non-futility hypothesis: A relative risk of good outcome measured by the Glasgow Outcome Scale-Extended 6 months after injury of 2.0 is consistent with the results of this phase II study.

ELIGIBILITY:
Inclusion Criteria:

1. Non-penetrating traumatic brain injury
2. Requirement for intracranial pressure monitoring according to Guidelines for the Management of Severe TBI, as operationalized below:

   * GCS 3-8 (measured off sedatives or paralytics) with abnormal CT scan. If patient is intubated, motor GCS < 4 required.
   * If CT scan normal, motor GCS < 4 (measured off sedatives or paralytics)
   * Intoxication is not a reason for deferring ICP monitoring if above criteria are met.
   * If the patient has a witnessed seizure, wait 30 minutes to evaluate GCS.
3. Randomization and placement of monitors within 12 hours of injury.
4. Males and females Age 18-70 years, English or Spanish speaking patients.

Exclusion Criteria:

1. Specific clinical contraindications:

   * GCS motor score > 4 with normal CT scan
   * Bilaterally absent pupillary responses
2. Laboratory contraindications per safety considerations:

   Coagulopathy that makes insertion of parenchymal monitors contraindicated (Platelets < 50,000/mL, INR > 1.4) (Enrollment allowed if coagulopathy can be corrected before 12 hour post-injury deadline).
3. Pregnant females will be excluded. Blood test for pregnancy is a routine part of care in ED's. However, if not done, a urine or blood test will be done as a safety precaution after consent but prior to study treatment.
4. Monitoring with pBrO2 monitor prior to randomization.
5. Clinical, demographic and other characteristics that precludes appropriate diagnosis, treatment or follow-up in the trial.

   * Systemic sepsis at the time of screening
   * Refractory hypotension (SBP < 70 mm Hg for > 30 minutes)
   * Refractory systemic hypoxia (paO2 < 60 mm Hg on FiO2 < 0.5)
   * Evidence of premorbid disabling conditions that interfere with outcome assessment. These include diagnosis of Alzheimer's disease, Parkinson's disease, multiple sclerosis, spinal cord injury with deficits, history of stroke, brain tumors, chronic use of medication for disabling neurologic or psychiatric disorder, or history of suicide attempt within the past year.
   * Imminent death or current life-threatening disease
   * Prisoner
   * Individuals who hold religious beliefs against blood transfusion
   * Previous TBI hospitalization greater than 1 day
   * Patients who are unlikely to be available for follow-up interview, even by telephone. for example, patients who are homeless, illegal aliens, or live in foreign countries and those with whom future personal (including family) or telephone contact is unlikely.
6. Active drug or alcohol use or dependence that, in the opinion of the stie investigator, would interfere with follow-up.
7. Imminent death or current life-threatening disease
8. Inability or unwillingness of subject or legal guardian/representative to give written informed consent
9. Participation in other observational or interventional clinical trials is allowed as long as the PI of each study agree ahead of time to allow co-enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2009-10; Primary Completion 2014-03 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of Miami/Jackson Memorial Hospital, Miami, Florida
  - Duke University, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Washington/Harborview Medical Center, Seattle, Washington

REFERENCES:
- [Result] Okonkwo DO, Shutter LA, Moore C, Temkin NR, Puccio AM, Madden CJ, Andaluz N, Chesnut RM, Bullock MR, Grant GA, McGregor J, Weaver M, Jallo J, LeRoux PD, Moberg D, Barber J, Lazaridis C, Diaz-Arrastia RR. Brain Oxygen Optimization in Severe Traumatic Brain Injury Phase-II: A Phase II Randomized Trial. Crit Care Med. 2017 Nov;45(11):1907-1914. doi: 10.1097/CCM.0000000000002619. PMID 29028696

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with severe TBI who required ICP monitoring were screened at 10 Level 1 trauma centers . Patients admitted with an initial GCS greater than 8 who deteriorated neurologically (within 48 hr of injury) from a presumptive could also be enrolled provided randomization and ICP monitor placement occurred within 12 hours of deterioration.
Period: Overall Study
Arm/Group | pBrO2 and ICP Management | ICP Management
Started | 59 | 63
Completed | 57 | 62
Not Completed | 2 | 1
Not completed — Technically inadequate PbtO2 recordings | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | pBrO2 and ICP Management | ICP Management | Total
Number analyzed (Participants) | 57 | 62 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 62 | 119
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (17.2) | 36.2 (17.5) | 37.0 (17.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 27
  Male | 46 | 46 | 92
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 47 | 53 | 100
  Black | 9 | 11 | 20
  Other | 2 | 2 | 4
  Unknown | 3 | 0 | 3
Injury Type--Closed Head Injury [Count of Participants; unit: Participants] | 56 | 62 | 118
Glasgow Come Scale-Motor [Mean (Standard Deviation); unit: units on a scale] — Glasgow Coma Scale is an ordinal scale measuring coma severity. Scale ranges from 3 (severe coma) to 15 (awake, alert, following commands), thus lower is worse, higher is better.
  units on a scale | 3.6 (1.5) | 3.7 (1.5) | 3.7 (1.5)
Craniectomy [Count of Participants; unit: Participants] | 12 | 18 | 30

OUTCOME MEASURES:

1. Primary Outcome: Fraction of Time That Brain Oxygen Levels Are Below the Critical Threshold of 20 mm Hg .
Description: Proportion of time PbtO2 below 20 mm Hg
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: Proportion
Arm/Group | pBrO2 and ICP Management | ICP Management
Number analyzed (Participants) | 57 | 62
Proportion | 0.15 (0.21) | 0.44 (0.31)

2. Secondary Outcome: Total Number Participants With Adverse Events Associated With PbtO2 Monitoring.
Description: Total number participants with PbtO2 directed intervention-related Serious Adverse Events
Time Frame: 5 days
Measure: Number; unit: participants
Arm/Group | pBrO2 and ICP Management | ICP Management
Number analyzed (Participants) | 57 | 62
participants
  Cardiovascular SAEs | 9 | 8
  Gastro-intestinal SAEs | 1 | 1
  Neurological SAEs | 5 | 10
  Respiratory SEAs | 4 | 1
  Other SAEs | 8 | 17
  Death Following withdrawal of medical care | 8 | 14

3. Secondary Outcome: Adherence to PbtO2 and ICP-directed Treatment Protocol
Description: Number of protocol deviations and violations for ICP/PbtO2 group and ICP only group.
  The unit of measure for this outcome is number of events, where an event can be either a deviation or a violation.
Time Frame: 5 days
Measure: Number; unit: Events (sum of deviations & violations)
Arm/Group | pBrO2 and ICP Management | ICP Management
Number analyzed (Participants) | 57 | 62
Events (sum of deviations & violations)
  Deviation: ICP 20-25 for > 30 min w/o Rx | 95 | 71
  Deviation: PbtO2 15-19 for > 30 min w/o Rx | 24 | 0
  Violation: ICP > 25 for > 30 min w/o Rx | 7 | 14
  Violation: PbtO2 < 15 for > 30 min w/o Rx | 17 | 0

4. Secondary Outcome: Relative Risk of Good Outcome of ICP/PbtO2 Group Compared to ICP Only Group.
Description: Dichotomized Glagow Outcome Score-Extended:
  GOSE 1-4 = Poor Outcome GOSE 5-8 = Good Outcome GOSE is a 8-point scale, with 1 = death, 8 = full recovery.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | pBrO2 and ICP Management | ICP Management
Number analyzed (Participants) | 57 | 62
participants
  GOSE 1 | 13 | 18
  GOSE 2 | 1 | 2
  GOSE 3 | 7 | 5
  GOSE 4 | 10 | 12
  GOSE 5 | 4 | 4
  GOSE 6 | 5 | 5
  GOSE 7 | 6 | 4
  GOSE 8 | 7 | 2

ADVERSE EVENTS:
Arm/Group | pBrO2 and ICP Management | ICP Management
All-Cause Mortality (participants affected / at risk) | 13/57 | 18/62
Serious Adverse Events (participants affected / at risk) | 27/57 | 34/62
Other Adverse Events (participants affected / at risk) | 48/57 | 55/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | pBrO2 and ICP Management (N=57) | ICP Management (N=62)
Cardiovascular (Cardiac disorders) | 9 (9) | 5 (5)
Pulmonary (General disorders) | 4 (4) | 1 (1)
Gastro-intestinal (Gastrointestinal disorders) | 1 (1) | 1 (1)
Neurological (Nervous system disorders) | 5 (5) | 10 (10)
Other (General disorders) | 8 (8) | 17 (17)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | pBrO2 and ICP Management (N=57) | ICP Management (N=62)
Other (General disorders) | 48 (48) | 55 (55)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No